CLINICAL TRIAL: NCT00385801
Title: A Double-Blind, Placebo-Controlled Study of the Effects of Risperdal Consta on Brain Reward Circuitry, Craving and Cocaine Use in Active Cocaine Dependence
Brief Title: Study of the Effects of Risperdal Consta on Brain Reward Circuitry Function, Craving and Cocaine Use in Active Cocaine Dependence
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Janssen, LP (Industry)
Responsible Party: Principal Investigator, A. Eden Evins, PI, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: RIS-EMR-4021
Record Dates: First submitted 2006-10-06; First posted 2006-10-11 (Estimated); Results first posted 2017-04-28 (Actual); Last update posted 2017-04-28 (Actual); Status verified 2017-03

CONDITIONS: Cocaine Dependence
Keywords: cocaine; dependence; risperidal; MRI
MeSH Terms: conditions — Cocaine-Related Disorders | interventions — Risperidone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator

ARMS (2):
- Placebo (Placebo Comparator): Identical placebo tablets and injections
  Interventions: Drug: Placebo
- risperidone consta (Active Comparator): Risperidone 1-2 mg tablets and Risperidone 25 mg injections
  Interventions: Drug: Risperidone

INTERVENTIONS:
Drug: Risperidone
  Arms: risperidone consta
Drug: Placebo
  Arms: Placebo

SUMMARY:
The purpose of this study is to examine the effects of the administration of Risperidal-Consta on the brain's reward circuitry using Magnetic resonance Imaging (MRI), behavioral tests and measuring cocaine craving and use among people with active cocaine dependence.

ELIGIBILITY:
Inclusion Criteria:

* current cocaine dependence who use cocaine at least every 2 weeks
* Non-treatment seekers who intend to continue using cocaine
* Male 18-60 years of age
* Potential participants must be literate in the English language, and be able to understand and complete rating scales and questionnaires accurately
* Able to provide informed consent
* Potential participants must be able to identify at least one "locator" person to assist in tracking the participant for follow-up assessments

Exclusion Criteria:

* Other current substance dependence requiring immediate detoxification
* Diagnosis of schizophrenia, bipolar disorder, current major depressive disorder
* Currently suicidal or at high risk for suicide in the judgment of the investigator
* Carrying a medical device incompatible with MRI (e.g., metal implants such as surgical clips or pacemakers and extensive dental work such as bridges) or suffering from significant claustrophobia that would make MRI unfeasible.
* Size incompatible with MRI procedures
* Serious medical illness including HIV-1 infection
* Hepatitis C + titer with liver enzymes more than 2x normal or a Mini-Mental Status Exam Score of <25/30
* Insulin dependent diabetes mellitus (IDDM) or non- insulin dependent diabetes mellitus (NIDDM) and abnormal Hemoglobin A1C
* Severe hepatic or renal impairment
* History of seizure disorder, delirium, dementia, or mental disorders due to general medical conditions
* History of head trauma or stroke with lasting neurological sequelae
* Tardive dyskinesia, extrapyramidal movement disorder, Parkinson's Disease or history of Neuroleptic Malignant Syndrome
* Clinical or laboratory evidence of uncontrolled hypothyroidism/hyperthyroidism
* Orthostatic hypotension, defined as a decrease of at > 10 mm Hg in systolic blood pressure and/or an increase in heart rate of > 20 beats per minute, measured one minute following transition from a supine to a standing position.
* History of allergy or hypersensitivity to Risperidone
* Treatment with: Neuroleptics, Antidepressants, Antiarrhythmics, Carbamazepine, Phenytoin, Valproate, Rifampin, Phenobarbital, Levodopa and other dopamine agonists, Fluoxetine, Interferon, Propylthiouracil, Methimazole, Opiates.
* Treatment within 30 days prior to screening with an investigational drug or medication with the potential to influence cocaine use outcomes

Ages: 18 Years to 60 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 31 (Actual)
Dates: Start 2005-09; Primary Completion 2010-09 (Actual); Study Completion 2010-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Eden A Evins, MD MPH, Principal Investigator — Massachusetts General Hospital
Locations (1):
- MGH Addiction Research Program, Boston, Massachusetts, United States

REFERENCES:
- [Derived] Loebl T, Angarita GA, Pachas GN, Huang KL, Lee SH, Nino J, Logvinenko T, Culhane MA, Evins AE. A randomized, double-blind, placebo-controlled trial of long-acting risperidone in cocaine-dependent men. J Clin Psychiatry. 2008 Mar;69(3):480-6. doi: 10.4088/jcp.v69n0321. PMID 18294021

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from October 2005 to September 2006 via advertisement in local press
Pre-assignment Details: After baseline evaluation participants began treatment with oral risperidone, 1 mg per day the first week and 2 mg per day for the next 3 weeks. Electrocardiograms were repeated after 1 and 2 weeks of risperidone use. Participants with corrected QT interval (QTc) prolongation greater than 470 milliseconds at either of these occasions were excluded
Period: Overall Study
Arm/Group | Placebo | Risperidone Consta
Started | 15 | 16
Completed | 6 | 8
Not Completed | 9 | 8

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Risperidone Consta | Total
Number analyzed (Participants) | 15 | 16 | 31
Age, Continuous [Mean (Standard Deviation); unit: years] | 42.4 (6.4) | 44.1 (5.9) | 43 (6.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 15 | 16 | 31

OUTCOME MEASURES:

1. Primary Outcome: Functional MRI Activation Patterns in the Nucleus Accumbens and Amygdala in Response to Cocaine Cues
Description: Measure of Dispersion/Precision not calculated, and raw data are no longer available
Time Frame: 12 weeks
Population: Measure of Dispersion/Precision not calculated, and raw data are no longer available
Arm/Group | Placebo | Risperidone Consta
Number analyzed (Participants) | 0 | 0

2. Primary Outcome: Cocaine Use by Quantitative Urine Samples
Description: After randomization, participants provided urine samples every week for the first 3 weeks and then every 2 weeks for 8 weeks, up to 7 samples per participant. The average visits with cocaine negative urine samples per participant are reported below
Time Frame: 12 weeks
Population: Mean number of visits at which participants submitted urine samples with undetectable urine benzoylecgonine (UBE)
Measure: Mean (Standard Deviation); unit: visit with negative UBE
Arm/Group | Placebo | Risperidone Consta
Number analyzed (Participants) | 15 | 16
visit with negative UBE | 1.81 (2.29) | 0.87 (1.8)

3. Secondary Outcome: Cocaine Craving
Description: The University of Minnesota Cocaine Craving Scale was performed to assess cocaine craving. The scale contains 1 continuous scale for intensity and 2 categorical scales for frequency and duration of craving episodes. The continuous scale for craving intensity ranges from 0 (no craving at all in the past week) to 10 (a great deal of craving in the past week)
Time Frame: 12 weeks
Population: Mixed model repeated measures analysis of variance was performed.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Risperidone: Risperidone 1-2 mg tablets and Risperidone 25 mg injections
Arm/Group | Placebo | Risperidone
Number analyzed (Participants) | 15 | 16
units on a scale | NA (NA) — Raw data to calculate the mean values and measure of Dispersion/Precision are no longer available | NA (NA) — Raw data to calculate the mean values and measure of Dispersion/Precision are no longer available
Statistical Analysis 1: Comparison: Placebo vs Risperidone; Intensity of craving; Test type: Superiority or Other; p = 0.86, Mixed Models Analysis — The effect of treatment on intensity of craving was assessed and the threshold for statistical significance was p < 0.05; F=0.03

4. Secondary Outcome: Amygdala Volume by MRI
Description: Measure of Dispersion/Precision not calculated, and raw data are no longer available
Time Frame: 12 weeks
Population: Measure of Dispersion/Precision not calculated, and raw data are no longer available
Arm/Group | Placebo | Risperidone Consta
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Adverse event data was collected at every visit
Arm/Group | Placebo | Risperidone Consta
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/16
Other Adverse Events (participants affected / at risk) | 7/15 | 13/16
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=15) | Risperidone Consta (N=16)
Increased appetite (General disorders) | 0 | 3
Common cold (Respiratory, thoracic and mediastinal disorders) | 0 | 4
Sexual dysfunction (Reproductive system and breast disorders) | 1 | 4
Insomnia (General disorders) | 0 | 2
Dizziness (General disorders) | 2 | 3
Dry mouth (General disorders) | 4 | 6
Rhinorrhea (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Sore throat (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Dyspepsia (Gastrointestinal disorders) | 3 | 2
Fatigue (General disorders) | 3 | 9
Somnolence (General disorders) | 2 | 9
Depression (Psychiatric disorders) | 2 | 2
Rash (Skin and subcutaneous tissue disorders) | 2 | 2
Increased thirst (General disorders) | 4 | 4
Muscle rigidity, twitches (Nervous system disorders) | 1 | 4
Increased urination (General disorders) | 0 | 2
Fever (General disorders) | 0 | 2
Parasthesia, hypoesthesia (Nervous system disorders) | 2 | 2
Akathisia (Nervous system disorders) | 0 | 2
Tardive dyskinesia (Nervous system disorders) | 0 | 1
Other (General disorders) | 3 | 7

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No